CLINICAL TRIAL: NCT00874679
Title: REal-Life Perception of Efficacy, Attitude, Satisfaction and Safety of Levitra® Therapy
Brief Title: REPEAT - Real-Life Perception of Efficacy, Attitude, Satisfaction and Safety of Levitra Therapy
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Other Study IDs: 12805; REPEAT (Other: Company Internal); LV0602 (Other: Company Internal); 12942 - LV0602KR (Other: Company Internal); 12975 - LV0602HR (Other: Company Internal); 12976 - LV0602CN (Other: Company Internal); 12977 - LV0602SG (Other: Company Internal); 13047 - LV0602SE (Other: Company Internal); 13048 - LV0602ZA (Other: Company Internal); 13067 - LV0602HU (Other: Company Internal); 13093 - LV0602MY (Other: Company Internal); 13112 - LV0602ID (Other: Company Internal); 13208 - LV0602TH (Other: Company Internal); 13416 - LV0602ES (Other: Company Internal); 13417 - LV0602SA (Other: Company Internal); 13600 - LV0602PL (Other: Company Internal); 14525 - LV0602FR (Other: Company Internal)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Patients with diagnosis of erectile dysfunction who get vardenafil in routine treatment

SUMMARY:
The aim of this prospective, non-interventional post-marketing surveillance study is to obtain data on safety and efficacy of Levitra in routine treatment of erectile dysfunction. Furthermore, the data collection particularly focuses on the experience of the patient and his satisfaction with the treatment. Treatment naive patients as well as pre-treated patients will be included in the study.The maximum observation period per patient is 12 months.Besides the physician's documentation, the patient should fill out a questionnaire at every visit. The questionnaires will be handed out and collected by the physician. Furthermore, an additional questionnaire for the patient's partner can be distributed at each visit in case the partner is willing to participate.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with diagnosis of erectile dysfunction, decision taken by the investigator to prescribe Vardenafil.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information. All contraindications listed in the local product information are applicable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of erectile dysfunction who get vardenafil in routine treatment
Sampling Method: Non-Probability Sample
Enrollment: 7293 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Physician's assessment of safety (incidence of adverse events) | During observation period

SECONDARY OUTCOMES:
Severity of ED symptoms | End of study
General quality of partnership as assessed by patient | Initial visit and after 3, 6, 9 and 12 months
General quality of partnership as assessed by partner | Initial visit and after 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Many Locations, China
- Many Locations, Croatia
- Many Locations, France
- Many Locations, Germany
- Many Locations, Hungary
- Many Locations, Indonesia
- Many Locations, Malaysia
- Many Locations, Poland
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, South Africa
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Thailand